CLINICAL TRIAL: NCT02348424
Title: Phase 1 Open Label Trial of the Safety, Tolerability, and Genitourinary and Pharyngeal Pharmacokinetics of Solithromycin
Brief Title: Genitourinary and Pharyngeal Pharmacokinetics of Solithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0069; HHSN272201500007I
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2017-04-05

CONDITIONS: Gonorrhoea
Keywords: genitourinary; Neisseriaceae; pharyngeal; Solithromycin
MeSH Terms: conditions — Gonorrhea | interventions — solithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female solithromycin (Experimental): 14 females will receive a single 1000mg dose of solithromycin after a 12 hour overnight fast (water permitted) administered orally.
  Interventions: Drug: Solithromycin
- Male solithromycin (Experimental): 14 males will receive a single 1000mg dose of solithromycin after a 12 hour overnight fast (water permitted) administered orally.
  Interventions: Drug: Solithromycin

INTERVENTIONS:
Drug: Solithromycin — Cohorts 1 and 2 will receive a single 1000mg dose of solithromycin after a 12 hour overnight fast (water permitted). Solithromycin is a fluoroketolide antibiotic under investigation for oral and parenteral use and will be administered orally.

SUMMARY:
This is an open-label Phase I study of plasma, genitourinary, rectal, and pharyngeal pharmacokinetics of a single 1000mg oral dose of solithromycin. Study Objectives: The primary objective is to determine the pharmacokinetics of solithromycin in plasma, vaginal, cervical, seminal, rectal, and pharyngeal fluid samples after a single 1000mg oral dose.

DETAILED DESCRIPTION:
This is an open-label Phase I study of plasma, genitourinary, rectal, and pharyngeal pharmacokinetics of a single 1000mg oral dose of solithromycin. A total of 28 subjects (14 male, 14 female) will be enrolled and will receive a single 1000mg dose of solithromycin after a 12 hour overnight fast (water permitted). Solithromycin is a fluoroketolide antibiotic under investigation for oral and parenteral use and will be administered orally. The study duration is approximately 18 months. Study Objectives: The primary objective is to determine the pharmacokinetics of solithromycin in plasma, vaginal, cervical, seminal, rectal, and pharyngeal fluid samples after a single 1000mg oral dose. The secondary objective is to determine the safety and tolerability of a single 1000 mg oral dose of solithromycin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and non-pregnant female subjects between 18 and 45 years of age (inclusive) -Body Mass Index (BMI) between 18 and 35 kg/m2 (inclusive) -Female sexually active subjects of must use one of the following acceptable birth control methods beginning 30 days prior to dosing and through 7 days post-dose: * Abstinence * Surgical sterilization * Hormonal contraceptives other than those inserted into the vagina (e.g. NuvaRing, intrauterine devices) -Male sexually active subjects must use one of the following acceptable birth control methods from 7 days prior to dosing through 7 days after dosing: * Abstinence * Surgical sterilization -Male subjects must agree not to donate sperm for 30 days after the solithromycin dose -Willingness and ability to provide written informed consent -Willingness and ability to adhere to the lifestyle guideline restrictions outlined in the protocol -Willingness and ability to participate in all study visits as required by the protocol, including optional overnight stays or returning to the unit on Days 1, 2, and 3.

Exclusion Criteria:

-Evidence or history of clinically significant disease or current infection. --oncologic, pulmonary, hepatic, gastrointestinal, cardiovascular, hematologic, metabolic, neurologic, immunologic, nephrologic, endocrine, or psychiatric disease -History of systemic (oral or parenteral) antibiotic use within two weeks prior to administration of study drug -Any condition possibly affecting drug absorption (e.g. status post gastrectomy) -History of post-antibiotic colitis within three months prior to screening -ECG with QTc > 450msec as corrected by the Fridericia formula for both males and females, or abnormal, clinically significant finding as reported by the overreading board certified cardiologist -Blood pressure readings >140 mmHg (systolic) or >90 mm/Hg (diastolic) -Participation in another research study or receipt of an investigational agent within 30 days of administration of the study drug * Investigational agent may include vaccine, drug, biologic, device, blood product, or medication. -Use of spermicide, an intrauterine device (IUD), diaphragm, and/or vaginally inserted hormonal contraceptive (e.g. NuvaRing) seven days prior to dosing -Treatment with any CYP3A4 enzyme altering drugs, except hormonal contraceptives or topical medications, within 14 days prior to treatment with study drug: --Use of systemic prescription drugs, vitamins, or herbal supplements, which in the opinion of the investigator may interfere with solithromycin metabolism via CYP3A4, within 14 days prior to administration of the study drug including, but not limited to * Concomitant use of drugs known to prolong the QT interval including class 1a (quinidine, procainamide) or Class III (amiodarone, sotalol), or antiarrythmics * Concomitant use of drugs, food, or herbal products known to be moderate to potent inhibitors of CYP3A4 isozymes: oral antifungal agents (e.g. ketoconazole, itraconazole, posaconazole, fluconazole and voriconazole); human immunodeficiency virus (HIV) protease inhibitors (e.g. ritonavir and saquinavir), hepatitis C virus (HCV) protease inhibitors (e.g. boceprevir and telaprevir), nefazodone, fluvoxamine, conivaptan, diltiazem, verapamil, aprepitant, ticlopidine, crizotinib, imatinib; grapefruit or grapefruit juice. * Any use within the prior 7 days of drugs or herbal products known to be moderate to potent inducers of CYP3A4 isozymes: St. John's Wort, rifampin, rifabutin, anti-convulsants (e.g. phenobarbital, carbamazepine, phenytoin, rufinamide), modafinil, armodafinil, etraverine, efavirenz, bosentan. * Required current use of drugs with narrow therapeutic indices that are principally metabolized by CYP3A4 or transported by P-glycoprotein (Pgp), for which a drug interaction with solithromycin could result in higher and possibly unsafe exposures to these drugs: e.g. the P-gp substrates digoxin or colchicine and the CYP3A4 substrates alfentanil, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, fentanyl, midazolam, pimozide, quinidine, sirolimus, tacrolimus, everolimus, and terfenadine. * Use of any non-prescription medications, vitamins, or dietary supplements , unless prior approval is granted by the investigator * Consumption of Seville oranges or products containing Seville orange components, grapefruit, or grapefruit juice within 14 days of administration of the study drug -Positive serum pregnancy test or breast feeding during the study -Positive test for human immunodeficiency virus (HIV-1), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibodies -Positive urine drug screen at Screening or Enrollment (Day -1) (marijuana, cocaine metabolite, amphetamines, opiates, phencyc lidine, methadone, barbiturates, and/or benzodiazepines) -Positive breathalyzer test for alcohol -Positive STI screen * GC, CT, syphilis, or trichomoniasis, symptomatic bacterial vaginosis (assessed by Amsel criteria), or vaginal discharge consistent with candidiasis (assessed by potassium hydroxide wet preparation) -History of clinically significant intolerance or hypersensitivity to macrolide antibiotics (as determined by the investigator) or any of the excipients in the solithromycin capsules. * Clinically significant intolerance is defined as severe nausea or vomiting after a standard dose. Note that mild nausea is common after macrolide administration and a prior history would not be a contraindication. * Likelihood of requiring treatment during the study with drugs not permitted by the protocol -Blood donation or other significant blood loss (as determined by the Investigator) within 56 days of screening -Plasma donation within seven days of screening -Laboratory values outside the eligibility ranges in the protocol (See protocol page 23 and Appendix C) for serum. -Laboratory values outside the eligibility ranges in the protocol (See protocol page 23 and Appendix C) for urinalysis. -Uncontrolled intercurrent illness (i.e. active infection) or fever (oral temperature >/=100.4 degrees Fahrenheit or >/= 38 degrees Celsius). -Known or suspected significant underlying illness including but not limited to, clinically significant liver disease, diabetes mellitus, or kidney impairment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics of solithromycin will be assessed by measurement of solithromycin levels in plasma, vaginal, cervical, seminal, rectal, and pharyngeal fluid samples at multiple time points after drug administration. | Day 1 to Day 3

SECONDARY OUTCOMES:
The safety and tolerability of a single 1000mg oral dose of solithromycin will be assessed by comparing ECGs to baseline ECGs | Day 1 to Day 7
The safety and tolerability of a single 1000mg oral dose of solithromycin will be assessed by laboratory analysis. | Day 1 to Day 7
The safety and tolerability of a single 1000mg oral dose of solithromycin will be assessed by reported adverse effects | Day 1 to Day 7
The safety and tolerability of a single 1000mg oral dose of solithromycin will be assessed by rotine vital signs | Day 1 to Day 7
The safety and tolerability of a single 1000mg oral dose of solithromycin will be assessed by routine physical exams | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland, United States